CLINICAL TRIAL: NCT01380639
Title: Effects of Vibration Training During a Three-week Rehabilitation on Exercise Capacity in Chronic Obstructive Pulmonary Disease (COPD) III/IV-Patients
Brief Title: Effects of Vibration Training on Exercise Capacity in COPD-patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, MD, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGL-Ga-6MGT-0810
Record Dates: First submitted 2011-04-01; First posted 2011-06-27 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD III/IV; 6-Minutes-Walking-Distance; Vibration training; Galileo; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation with vibration training (Experimental)
  Interventions: Other: whole body vibration training
- Rehabilitation without vibration training (No Intervention)

INTERVENTIONS:
Other: whole body vibration training — performing squats for 3x3 minutes while using vibration platform three times a week
  Arms: Rehabilitation with vibration training

SUMMARY:
The aim of this study is to investigate the exercise capacity in COPD-patients performing a vibration training additional to a standard three-week rehabilitation program in comparison to patients performing merely a rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Chronic obstructive pulmonary disease III/IV

Exclusion Criteria:

* Severe exacerbations in the last 4 weeks prior to begin of study (definition of exacerbation: symptoms on more than 3 days with a relevant change in drug therapy (cortisone, antibiotics))
* Severe disease other than COPD, that could influence the results of the study
* Abuse of alcohol or drugs
* Simultaneously participation in another study
* Tachypnea (>30/min)
* Severe exacerbation during rehabilitation
* Cardiac insufficiency (NYHA IV)
* Myocardial infarction during the last 6 weeks
* Mental-health problem
* Pregnancy
* Known HIV-infection
* Slipped disk
* Acute discopathy
* Acute thrombosis
* Implants in trained regions of the body (lower extremities)
* Acute inflammation of the locomotor system, active arthrosis or rheumatoid arthritis
* Acute tendinopathy in trained regions of the body
* Acute hernia
* Fresh fractures, wounds or scars in trained regions of the body
* Gallstones or stones in the urinary tract collection system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinikum Berchtesgadener Land, Schönau am Königssee, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment of patients is meant for the number of study completers without drop out patients (n=10).
Groups:
- Rehabilitation With Vibration Training: whole body vibration training : performing squats for 3x3 minutes while using vibration platform three times a week
Period: Overall Study
Arm/Group | Rehabilitation With Vibration Training | Rehabilitation Without Vibration Training
Started | 42 | 40
Completed | 36 | 36
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rehabilitation With Vibration Training | Rehabilitation Without Vibration Training | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 19 | 41
  >=65 years | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11) | 65 (7) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 19 | 21 | 40
Region of Enrollment [Number; unit: participants]
  Germany | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: 6-Minute-Walking-Distance
Description: Change in 6-minute-walking-distance from baseline to day 19
Time Frame: day 1, day 19
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Rehabilitation With Vibration Training | Rehabilitation Without Vibration Training
Number analyzed (Participants) | 36 | 36
m | 64 (59) | 37 (52)

2. Secondary Outcome: Body Composition
Description: Change in body composition from baseline to day 19
Time Frame: day 1 and 19
Reporting Status: Not Posted

3. Secondary Outcome: Isometric Maximum Handgrip Force
Description: change in isometric max. handgrip force from baseline to day 19
Time Frame: day 1, day 19
Reporting Status: Not Posted

4. Secondary Outcome: BODE-Score
Description: Change in Bode-Score from baseline to day 19
Time Frame: day 1, day 19
Reporting Status: Not Posted

5. Secondary Outcome: Lung Function
Time Frame: day 1
Reporting Status: Not Posted

6. Secondary Outcome: Arterial Blood Gas
Time Frame: day 1
Reporting Status: Not Posted

7. Secondary Outcome: Brain Natruretic Peptide (BNP)
Description: change in BNP from baseline to day 19
Time Frame: day 1, day 19
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 weeks during the study period
Groups:
- Rehabilitation Without Vibration Training: control intervention : performing squats for 3x3 minutes on the floor three times a week
Arm/Group | Rehabilitation With Vibration Training | Rehabilitation Without Vibration Training
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes